CLINICAL TRIAL: NCT06574776
Title: Prevalence and Associated Mortality of Infections by Multidrug-Resistant Organisms in Adults Intensive Care Units in Argentina (PREV-AR)
Brief Title: Prevalence and Associated Mortality of Infections by Multidrug-Resistant Organisms in Adults Intensive Care Units
Acronym: PREV-AR
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, MARIA INES STANELONI, MD, Hospital Italiano de Buenos Aires
Other Study IDs: PREV-AR
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Infectious Disease
Keywords: antimicrobial resistance; critical care
MeSH Terms: conditions — Communicable Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A single cohort: It is a study with a single cohort.
  Interventions: Other: Observation and collecting data

INTERVENTIONS:
Other: Observation and collecting data — In that single cohort we will collect data on MDRO infection and colonization prevalence, clinical characteristics, infections, causative organisms and mortality.

SUMMARY:
Observational 24-hr point prevalence study with longitudinal follow-up at 164 ICUs in Argentina. All adult patients (aged ≥18 years) at a participating ICU on November 24-28, 2023 with 60- day follow-up, were included. Epidemiological variables, sites of infection, isolated microorganisms, CPE colonisation, and hospital characteristics were collected. Main outcome measure was ICU mortality.

DETAILED DESCRIPTION:
Methods Study design PREVAR (PREValence of infection by MDR-microorganisms in ARgentina) was a national, cross-sectional, 24-hour multicentre study designed and conducted by SADI and SATI in Argentine ICUs.

Participants Sites were recruited to participate via announcements in national meetings, official societies' websites, social media, three online meetings explaining the project, and emails to all society members. Hospitals were registered on a secure website, where local investigators recorded main site characteristics in an electronic form.

Patient data were entered in an electronic case report form (CRF) using the Research Electronic Data Capture (REDCap) database (appendix 2). Local researchers were trained through online meetings on how to fill out the CRF. A centralized data center was responsible for managing the database and monitoring data quality in close contact with local researchers to minimize the occurrence of missing data. A dedicated email address was created to streamline communication.

Individual patient data were anonymised by assigning a numerical code to each case and recorded in order of admission.

Each local institutional review board approved the study and established the requirement for informed consent.

The PREVAR study protocol is available in appendix 3. All adult patients, 18 years and older, present on a participating ICU on the study day during the 24-h period (beginning at 8.00 a.m.) were included. The exact date could be selected from November 24-28, 2023, to ease logistics for individual sites. The patients present on day 1 in the ICU were available for inclusion in the cohort, which was then followed for mortality. There were no exclusion criteria.

Procedures The CRF included baseline and demographic characteristics of the study participants: date of hospital and ICU admission, age, gender, comorbid conditions, APACHE II and SOFA scores registered on admission; risk factors for MDRO infection during the previous six months, such as previous admission to a hospital, colonisation by Enterobacterales spp (only colonisation by CPE was measured, as it is the only type of colonisation usually monitored in Argentinian ICUs) and antibiotic utilization; type of admission (medical, elective or emergency surgery) was also collected. Data regarding colonisation by carbapenemase-producing Enterobacterales during the period occurring between hospital admission to enrollment was documented, whether colonisation had been detected in the hospital or in the ICU. SOFA score was also calculated on the day of enrollment.

Patient clinical status regarding infection was recorded by the treating physician according to the SEPSIS-3 definitions as: without infection, with infection but no sepsis, sepsis, and septic shock.10 In addition, infections were considered as definite (microbiologically confirmed), and probable or possible, according to the International Sepsis Forum definitions (ISF) for pneumonia, bloodstream infections (including infective endocarditis), intravascular catheter-related sepsis, intra-abdominal infections, urosepsis, and surgical wound infections. 11 In the cases where culture results were pending, categorisation was reviewed with the main investigators when the results were made available. Definitions of infection sites were those provided by the ISF. 11 Infections were registered as community-acquired, ICU-acquired, hospital non-ICU acquired, or as originating in long term care facilities.

According to microbiological findings, infections were recorded as MDRO or non-MDRO. MDRO's of interest were A.baumannii, difficult-to treat P. aeruginosa, carbapenemase-producing enterobacterales, extended spectrum β-lactamase producing microorganisms (ESBL), vancomycin-resistant enterococci, and methicillin-resistant S. aureus (MRSA) If available, further diagnostic methods were performed to further classified them as: KPC carbapenemase-producing enterobacterales (KPC), metallo-beta-lactamases (MBL), oxacillinases (OXA), extended spectrum β-lactamase (ESBL) producing organisms and AMPC beta-lactamases. The group of infections produced by non-MDRO for this study included infections by S.pneumoniae, S.pyogenes, S.aureus, E.Coli,, coagulase-negative Staphylococcus, Proteus sp., KES (Klebsiella-Enterobacter-Serratia-Citrobacter (KESC) group, C. difficile, and others.

The prescribed antimicrobial treatment was classified as empiric or targeted, according to the presence or not of positive cultures; for targeted treatment as adequate or inadequate, according to antimicrobial susceptibility testing; as utilizing novel or "old" antibiotics according to the European guidelines for the treatment of infections caused by multidrug-resistant Gram-negative bacilli 12; and as receiving Access, Watch and Reserve antibiotic groups according to the AWaRe WHO classification.) 13 Patients were followed until ICU discharge or death in the ICU.

Hospitals were classified as general or specialized, and as public or private. The number of total hospital beds were recorded as well as ICU beds, and the availability of certain relevant resources, such as infection control committee and antimicrobial stewardship program. Additionally, MDRO surveillance for infections and colonisation and how frequently it was performed (weekly, at ICU admission and/or before surgery) was detailed. Methods used to detect mechanisms of bacterial resistance were recorded as phenotypical, molecular or immunochromatographic.

The protocol of the study, the CRF and all the definitions appear in the Operations Manual (appendix 4).

Outcomes The main outcome measure was the prevalence of infection by MDRO. Secondary outcome measures were overall ICU mortality and its independent determinants, 28-day ICU mortality, determinants of infections by MDRO, prevalence of colonisation by CPE, and of infection in general, and ICU length of stay. Data was censored for 60 days.

Statistical analysis Prevalence was calculated as the number of infections caused by MDROs divided by the number of patients in the ICU on the day of the study.

Variables are reported as absolute numbers and percentages, or as medians and interquartile ranges (IQRs). Differences in recorded variables between patients with MDRO and non-MDRO infections, between survivors and non-survivors, and between patients with and without infection were analyzed using the χ² test or Fisher's exact test for categorical variables, and the t test or Wilcoxon rank-sum test for continuous variables, as appropriate.

To estimate the associations of patient characteristics, ICU organizational factors, and hospital characteristics with infection by MDRO and ICU mortality, a mixed-effects model was performed. These models have a hierarchical structure with patients (level 1) nested within hospitals (level 2). This nesting accounts for the potential correlation of outcomes within the same hospital. Random Effects: Hospitals were treated as random effects to account for the potential correlation of outcomes within the same hospital and to capture variability between hospitals through random intercepts Fixed Effects: Patient characteristics and ICU organizational factors were included as fixed effects, as these are the primary predictors of interest.

Only variables with a P value <.20 in the bivariable analysis were introduced into the final model. The results for fixed effects are reported as odds ratios (ORs) with 95% confidence intervals (CIs). Random effects, or measures of variation, are reported as the variance, its standard error (SE), and the median OR. The statistical significance of covariates was determined using the likelihood ratio test.

All reported p values are two-sided, with a p value <0.05 considered statistically significant.

The funder of the study had no role in study design, data collection, data analysis, data interpretation, or writing of the report.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, 18 years and older, present on a participating ICU on the study day during the 24-h period (beginning at 8.00 a.m.) were included.

Exclusion Criteria:

* There were no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The exact date could be selected from November 24-28, 2023, to ease logistics for individual sites. The patients present on day 1 in the ICU were available for inclusion in the cohort, which was then followed for mortality.
Sampling Method: Non-Probability Sample
Enrollment: 1799 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
prevalence of infection by MDRO | All adult patients, 18 years and older, present on a participating ICU on the study day during the 24-h period (beginning at 8.00 a.m.) were included. The exact date could be selected from November 24-28, 2023.
  The main outcome measure was the prevalence of infection by MDRO.

SECONDARY OUTCOMES:
ICU mortality | 28 days
  28 days mortality and its independent determinants
prevalence of colonisation by MDRO | All adult patients, 18 years and older, present on a participating ICU on the study day during the 24-h period (beginning at 8.00 a.m.) were included. The exact date could be selected from November 24-28, 2023.
  prevalence of colonisation by multidrug resistant organisms
prevalence of infection in general | All adult patients, 18 years and older, present on a participating ICU on the study day during the 24-h period (beginning at 8.00 a.m.) were included. The exact date could be selected from November 24-28, 2023.
  prevalence of infection in general in the ICU on the study date

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Staneloni, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (7):
- Argentina (7):
  - Hospital Austral, Buenos Aires
  - Hospital de San Martin de La Plata, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Hospital Pirovano, Buenos Aires
  - Hospital Tornu, Buenos Aires
  - Sanatorio Las Lomas, Buenos Aires
  - Hospital de Clínicas Pte Nicolás Avellaneda, San Miguel de Tucumán

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cornistein W, Balasini C, Nuccetelli Y, Rodriguez VM, Cudmani N, Roca MV, Sadino G, Brizuela M, Fernandez A, Gonzalez S, Aguila D, Macchi A, Staneloni MI, Estenssoro E; Prevar Study Group. Prevalence and mortality associated with multidrug-resistant infections in adult intensive care units in Argentina (PREV-AR). Antimicrob Agents Chemother. 2025 Mar 5;69(3):e0142624. doi: 10.1128/aac.01426-24. Epub 2025 Jan 22. PMID 39840911